CLINICAL TRIAL: NCT00113581
Title: A Phase I Study to Determine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Three Doses of Humanised EGFR Antibody EMD 72000 in Combination With ECX in Patients With Advanced Oesophagogastric Adenocarcinoma
Brief Title: Safety Study of EMD 72000 in Combination With ECX (Epirubicin, Cisplatin and Capecitabine) in Oesophagogastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMD 72000-024
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: EMD 72000; matuzumab; Esophageal adenocarcinoma; Gastric adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — matuzumab

INTERVENTIONS:
Drug: EMD 72000 (matuzumab) + ECX

SUMMARY:
The main purpose of this study is to test the safety and tolerability and effectiveness of a new treatment, EMD 72000 (matuzumab), for advanced oesophagogastric cancer in combination with the chemotherapy regimen ECX (epirubicin, cisplatin and capecitabine).

In addition the study will look at pharmacokinetic (how the the body takes up the drug) and pharmacodynamic parameters (what the drug does in the body).

ELIGIBILITY:
Inclusion Criteria:

* Advanced, recurrent or metastatic gastric adenocarcinoma or adenocarcinoma of the lower third of the esophagus
* EGFR positive tumor
* KPS greater than 60
* Normal cardiac function
* Adequate liver and bone marrow function
* GFR greater than 60 ml/minute

Exclusion Criteria:

* Previous chemotherapy
* Uncontrolled angina pectoris, heart failure, clinically significant uncontrolled cardiac arrythmias
* Clinically significant ECG or cardiac history
* Radiotherapy or surgery within last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2002-10; Primary Completion 2006-05 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacodynamic parameters
Pharmacokinetic parameters
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Professor, Principal Investigator — The Royal Marsden Hospital, Sutton, UK
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom